CLINICAL TRIAL: NCT05328297
Title: A Randomized, Stratified, Double-blind, Placebo-Controlled Study to Investigate the Efficacy, Safety and Tolerability of JNJ-55308942 in Bipolar Depression
Brief Title: A Study of JNJ-55308942 in the Treatment of Bipolar Depression
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109116; 2021-004790-31 (EudraCT Number); 55308942BIP2001 (Other: Janssen Pharmaceutica N.V., Belgium)
Record Dates: First submitted 2022-04-11; First posted 2022-04-14 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Bipolar Disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — JNJ-55308942

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-55308942 (Experimental): Participants will receive a JNJ-55308942 capsule once daily for 6 weeks.
  Interventions: Drug: JNJ-55308942
- Placebo (Placebo Comparator): Participants will receive a matching placebo capsule once daily for 6 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-55308942 — JNJ-55308942 capsules will be administered orally.
  Arms: JNJ-55308942
Drug: Placebo — Matching placebo capsules will be administered orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of JNJ-55308942 compared to placebo on symptoms of depression in participants with bipolar disorder (BD) in a major depressive episode (MDE) at Week 6.

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnostic and statistical manual of mental disorders (5th edition) (DSM-5) diagnosis of bipolar disorder (BD) (Type I or II) without current psychotic features, as confirmed by the mini international neuropsychiatric interview (MINI)
* Medically stable on the basis of physical examination, medical history, and vital signs performed at screening. Any abnormalities must be consistent with the underlying illness in the study population. This determination must be recorded in the participant's source documents and initialed by the investigator
* Have a body mass index (BMI) between 18.0 and 35.0 kilograms per meter square (kg/m^2) inclusive (BMI = weight/height^2)
* A woman of childbearing potential (WOCBP) must have a negative highly sensitive serum pregnancy test (beta-human chorionic gonadotropin [beta-hCG]) at screening and a negative urine pregnancy test before the first dose of study intervention

Exclusion Criteria:

* Currently meets the DSM-5 criteria for Manic Episode (ME) on the MINI
* Received transcranial magnetic stimulation (TMS), any transcranial electrical stimulation, including transcranial direct current stimulation (tDCS), vagal nerve stimulation (VNS) and/or deep brain stimulation (DBS) within 6 weeks prior to randomization
* History of moderate to severe cannabis misuse according to DSM-5 criteria within 6 months before screening
* History of malignancy within 5 years before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator is considered cured with minimal risk of recurrence)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2024-05-17 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (44):
- United States (18):
  - UAB Huntsville Regional Medical Campus, Huntsville, Alabama
  - Preferred Research Partners, Little Rock, Arkansas
  - Synergy East, Lemon Grove, California
  - Collaborative NeuroScience Network, Torrance, California
  - Clinical Neuroscience Solutions Inc, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Psychiatric Medicine Associates LLC, Skokie, Illinois
  - Indiana University, Indianapolis, Indiana
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Richard H. Weisler, MD & Associates, Raleigh, North Carolina
  - Case Western Reserve School of Medicine, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Clinical NeuroScience Solutions Inc, Memphis, Tennessee
  - The University of Texas at Austin Department of Psychiatry, Dell Medical School, Austin, Texas
  - North Texas Clinical Trials, Fort Worth, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Northwest Clinical Research Center, Bellevue, Washington
- Canada (2):
  - The Medical Arts Health Research Group, West Vancouver, British Columbia
  - Chatham-Kent Clinical Trials Research Centre, Chatham, Ontario
- Poland (14):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku Klinika Psychiatrii, Bialystok
  - PROMENTE Sp. z o.o., Bydgoszcz
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Specjalistyczna Praktyka Lekarska Piotr Zalitacz, Gorlice
  - Centrum Medyczne Care Clinic Katowice, Katowice
  - Indywidualna Praktyka Lekarska Kinga Bobinska, Lodz
  - Filip Rybakowski Specjalistyczna Praktyka Lekarska, Poznan
  - Centrum Medyczne HCP Sp. z o.o. Osrodek Badan Klinicznych, Poznan
  - Samodzielny Publiczny Zespol Lecznictwa Psychiatrycznego w Siemianowicach Slaskich, Siemianowice Śląskie
  - Indywidualna Specjalistyczna Praktyka Lekarska Agnieszka Remlinger Molenda, Suchy Las
  - Szpital Nowowiejski Osrodek Badan Klinicznych, Warsaw
  - Instytut Psychiatrii I Neurologii, Warsaw
  - Przychodnia Lekarsko-Psychologiczna Persona, Wroclaw
  - Ginemedica Sp. z o.o., Wroclaw
- Spain (10):
  - Hosp. Del Mar, Barcelona
  - Institucion Hosp Hestia Palau, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Centro Salud Mental La Eria, Oviedo
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. El Bierzo, Ponferrada
  - Hosp. Univ. I Politecni La Fe, Valencia
  - Hosp. Alvaro Cunqueiro, Vigo
  - Hosp. Psiquiatrico Alava, Vitoria-Gasteiz

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

RESULTS

PARTICIPANT FLOW:
Groups:
- JNJ-55308942: During double-blind (DB) treatment phase, participants received JNJ-55308942 capsule, orally once daily from Day 1 (Week 0) up to 6 weeks. Participants were then followed up for up to 2 weeks after their last dose (up to Day 56).
- Placebo: During DB treatment phase, participants received placebo capsule (matching to JNJ-55308942), orally once daily from Day 1 (Week 0) up to 6 weeks. Participants were then followed up for up to 2 weeks after their last dose (up to Day 56).
Period: Overall Study
Arm/Group | JNJ-55308942 | Placebo
Started | 55 | 61
Treated (Safety Analysis Set) | 54 (Included one participant from placebo arm who received JNJ-55308942 erroneously.) | 60
Completed | 42 | 50
Not Completed | 13 | 11
Not completed — Adverse Event | 5 | 7
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — Randomized but not treated | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all randomized participants who received at least 1 dose of study treatment in the double-blind (DB) treatment phase.
Groups:
- Total: Total of all reporting groups
Arm/Group | JNJ-55308942 | Placebo | Total
Number analyzed (Participants) | 54 | 60 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.28 (13.603) | 40.18 (12.664) | 39.75 (13.067)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 33 | 71
  Male | 16 | 27 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 50 | 53 | 103
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 8 | 8 | 16
  White | 44 | 50 | 94
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 1 | 0 | 1
  Poland | 30 | 30 | 60
  Spain | 2 | 5 | 7
  United States | 21 | 25 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score up to Week 6
Description: Change from baseline in MADRS total score up to Week 6 were reported. MADRS was a clinician-rated scale designed to measure depression severity and detect changes due to antidepressant (AD) treatment. The MADRS evaluated reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The scale consisted of 10 items, each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms),with higher score indicating a more severe condition. The MADRS total score was the sum of scores from individual question items and it ranged from 0 to 60, with higher scores indicated more severe conditions. Negative change in MADRS total score indicated improvement.
Time Frame: From Baseline (Day 1) up to Week 6
Population: Full analysis set (FAS) included all randomized participants who received at least 1 dose of study intervention and had both the baseline and at least 1 postbaseline MADRS measurement.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 48 | 59
Units on a scale | -16.0 (10.43) | -15.4 (9.81)
Statistical Analysis 1: Comparison: JNJ-55308942 vs Placebo; Test type: Superiority; p = 0.438, Mixed Model for Repeated Measures (MMRM); Least Square Mean difference = -0.3, 80% CI 2-sided [-2.84 to 2.23], Standard Error of Mean 1.96

2. Secondary Outcome: Change From Baseline in Snaith-Hamilton Pleasure Scale (SHAPS) Total Score up to Week 6
Description: Change from baseline in SHAPS total score up to Week 6 were reported. The SHAPS was a reliable, valid, and unidimensional instrument used to assess hedonic capacity in adults with Major Depressive Disorder. It is a 14-item, self-report tool with a completion time below 5 minutes. Each of the items had a set of 4 response categories: 1 = definitely agree/strongly agree, 2 = agree, 3 = disagree, and 4 = strongly disagree. The SHAPS total score was the sum of the 14 item scores, which ranged from 14 to 56. A higher SHAPS total score indicated higher levels of current anhedonia. Negative changes in the SHAPS total score indicated improvement.
Time Frame: From Baseline (Day 1) up to Week 6
Population: FAS included all randomized participants who received at least 1 dose of study intervention and had both the baseline and at least 1 postbaseline MADRS measurement. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 42 | 50
Units on a scale | -8.2 (6.87) | -8.3 (8.69)

3. Secondary Outcome: Change From Baseline in MADRS Total Score up to Week 6 (Genetic Subgroup Analysis)
Description: Genetic subgroup analysis included participants with bipolar depression and who were with P2RX7 Gain of Function single nucleotide polymorphism (P2RX7 GoF SNP) mutation genotype: heterozygous or homozygous. MADRS was a clinician-rated scale designed to measure depression severity and detect changes due to AD treatment. The MADRS evaluated reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The scale consisted of 10 items, each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms),with higher score indicating a more severe condition. The MADRS total score was the sum of scores from individual question items and it ranged from 0 to 60, with higher scores indicated more severe conditions. Negative change in MADRS total score indicated improvement.
Time Frame: From Baseline (Day 1) up to Week 6
Population: FAS included all randomized participants who received at least 1 dose of study intervention and had both the baseline and at least 1 postbaseline MADRS measurement. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed at specified categories.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 42 | 50
Units on a scale
  P2RX7 GoF SNP mutation genotype: Heterozygous: number analyzed (Participants) | 31 | 34
  P2RX7 GoF SNP mutation genotype: Heterozygous | -15.2 (9.45) | -16.5 (10.22)
  P2RX7 GoF SNP mutation genotype: Homozygous: number analyzed (Participants) | 11 | 16
  P2RX7 GoF SNP mutation genotype: Homozygous | -18.2 (13.06) | -13.1 (8.75)

4. Secondary Outcome: Change From Baseline in MADRS Total Score up to Week 6 (Diagnosis Subgroup Analysis)
Description: Change from baseline in MADRS total score up to Week 6 (Diagnosis Subgroup Analysis) were reported. Diagnosis subgroup analysis included participants with bipolar type 1 or II. MADRS was a clinician-rated scale designed to measure depression severity and detect changes due to AD treatment. The MADRS evaluated reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The scale consisted of 10 items, each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms),with higher score indicating a more severe condition. The MADRS total score was the sum of scores from individual question items and it ranged from 0 to 60, with higher scores indicated more severe conditions. Negative change in MADRS total score indicated improvement.
Time Frame: From Baseline (Day 1) up to Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 42 | 50
Units on a scale
  Bipolar type I: number analyzed (Participants) | 33 | 37
  Bipolar type I | -15.5 (11.02) | -15.3 (10.06)
  Bipolar type II: number analyzed (Participants) | 9 | 13
  Bipolar type II | -17.7 (8.20) | -15.7 (9.47)

5. Secondary Outcome: Change From Baseline in MADRS Total Score up to Week 6 (Biomarker Subgroup Analysis)
Description: Biomarker subgroup analysis included specific (3-Marker Model [3MM]) biomarker profile: Yes or No. 3MM biomarker profile was defined as serum C-reactive protein >3 mg/Liter(L) and soluble interleukin-6 receptor >25 micrograms(mcg)/L or tumor necrosis factor >4 nanograms(ng)/L at baseline. MADRS was a clinician-rated scale designed to measure depression severity and detect changes due to AD treatment. MADRS evaluated reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. Scale consist of 10 items each of which was scored from 0(item not present or normal) to 6(severe or continuous presence of the symptoms),with higher score indicating a more severe condition. MADRS total score was sum of scores from individual question items, ranged from 0 to 60,with higher scores indicated more severe conditions. Negative change in MADRS total score indicated improvement.
Time Frame: From Baseline (Day 1) up to Week 6
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 42 | 49
Units on a scale
  3MM biomarker profile: Yes: number analyzed (Participants) | 11 | 22
  3MM biomarker profile: Yes | -12.5 (9.04) | -13.9 (10.77)
  3MM biomarker profile: No: number analyzed (Participants) | 31 | 27
  3MM biomarker profile: No | -17.2 (10.75) | -16.6 (9.17)

6. Secondary Outcome: Number of Participants With Treatment-emergent Clinically Important Abnormalities in Vital Signs
Description: Vital signs parameters included pulse rate (abnormally low [AL]: <50 beats per minute [bpm] and with >15 bpm decrease from baseline and abnormally high [AH]: >100 bpm and with >15 bpm increase from baseline), Systolic blood pressure (SBP) (AL: <90 millimeters of mercury [mmHg] and with >20 mmHg decrease from baseline and AH: >180 mmHg and with >20 mmHg increase from baseline), Diastolic blood pressure (DBP) (AL: <50 mmHg and with >15 mmHg decrease from baseline and AH: >105 mmHg and with >15 mmHg increase from baseline) , temperature (AL:<35.5 and AH:>37.5 degree Celsius [C]), respiratory rate (AH :>20 breaths per minute), and weight (AL: decrease from baseline >7% and AH: increase from baseline >7%). Weight was planned to analyzed at Weeks 6 and 8 only. Treatment-emergent concluded if postbaseline value was above/below upper/lower limit and baseline value was below/above the upper/lower limit.
Time Frame: Weeks 1, 2, 4, 6, and 8 (Follow-up/Early Withdrawal)
Population: Safety analysis set included all randomized participants who took at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 49 | 56
Participants
  Pulse (beats per minutes [bpm]): <50 bpm and with >15 bpm decrease from baseline: Week 1 | 0 [lower limit 9.04] | 0 [lower limit 10.77]
  Pulse (bpm): >100 bpm and with >15 bpm increase from baseline: Week 1 | 0 [lower limit 10.75] | 0 [lower limit 9.17]
  SBP (millimeters of mercury [mmHg]): <90 mmHg and with >20 mmHg decrease from baseline: Week 1 | 0 | 0
  SBP (mmHg): >180 mmHg and with >20 mmHg increase from baseline: Week 1 | 0 | 0
  DBP (mmHg): <50 mmHg and with >15 mmHg decrease from baseline : Week 1 | 0 | 0
  DBP (mmHg): >105 mmHg and with >15 mmHg increase from baseline: Week 1 | 0 | 0
  Temperature (degree Celsius [C]): <35.5 degree C: Week 1: number analyzed (Participants) | 46 | 56
  Temperature (degree Celsius [C]): <35.5 degree C: Week 1 | 0 | 0
  Temperature (degree C): >37.5 degree C: Week 1: number analyzed (Participants) | 46 | 56
  Temperature (degree C): >37.5 degree C: Week 1 | 0 | 0
  Respiratory Rate: >20 breaths per minute: Week 1 | 0 | 0
  Pulse: <50 bpm and with >15 bpm decrease from baseline: Week 2: number analyzed (Participants) | 45 | 56
  Pulse: <50 bpm and with >15 bpm decrease from baseline: Week 2 | 0 | 0
  Pulse: >100 bpm and with >15 bpm increase from baseline: Week 2: number analyzed (Participants) | 45 | 56
  Pulse: >100 bpm and with >15 bpm increase from baseline: Week 2 | 0 | 0
  SBP:<90 mmHg and with >20 mmHg decrease from baseline: Week 2: number analyzed (Participants) | 45 | 56
  SBP:<90 mmHg and with >20 mmHg decrease from baseline: Week 2 | 0 | 0
  SBP: >180 mmHg and with >20 mmHg increase from baseline: Week 2: number analyzed (Participants) | 45 | 56
  SBP: >180 mmHg and with >20 mmHg increase from baseline: Week 2 | 0 | 0
  DBP: <50 mmHg and with >15 mmHg decrease from baseline: Week 2: number analyzed (Participants) | 45 | 56
  DBP: <50 mmHg and with >15 mmHg decrease from baseline: Week 2 | 0 | 0
  DBP: >105 mmHg and with >15 mmHg increase from baseline: Week 2: number analyzed (Participants) | 45 | 56
  DBP: >105 mmHg and with >15 mmHg increase from baseline: Week 2 | 0 | 0
  Temperature (degree C): <35.5 degree C: Week 2: number analyzed (Participants) | 45 | 56
  Temperature (degree C): <35.5 degree C: Week 2 | 0 | 0
  Temperature (degree C): >37.5 degree C: Week 2: number analyzed (Participants) | 45 | 56
  Temperature (degree C): >37.5 degree C: Week 2 | 0 | 0
  Respiratory Rate: >20 breaths per minute: Week 2: number analyzed (Participants) | 45 | 56
  Respiratory Rate: >20 breaths per minute: Week 2 | 0 | 1
  Pulse (bpm): <50 bpm and with >15 bpm decrease from baseline: Week 4: number analyzed (Participants) | 44 | 50
  Pulse (bpm): <50 bpm and with >15 bpm decrease from baseline: Week 4 | 0 | 0
  Pulse (bpm): >100 bpm and with >15 bpm increase from baseline: Week 4: number analyzed (Participants) | 44 | 50
  Pulse (bpm): >100 bpm and with >15 bpm increase from baseline: Week 4 | 0 | 0
  SBP (mmHg): <90 mmHg and with >20 mmHg decrease from baseline: Week 4: number analyzed (Participants) | 44 | 50
  SBP (mmHg): <90 mmHg and with >20 mmHg decrease from baseline: Week 4 | 0 | 0
  SBP (mmHg): >180 mmHg and with >20 mmHg increase from baseline: Week 4: number analyzed (Participants) | 44 | 50
  SBP (mmHg): >180 mmHg and with >20 mmHg increase from baseline: Week 4 | 0 | 0
  DBP (mmHg): <50 mmHg and with >15 mmHg decrease from baseline: Week 4: number analyzed (Participants) | 44 | 50
  DBP (mmHg): <50 mmHg and with >15 mmHg decrease from baseline: Week 4 | 0 | 0
  DBP (mmHg): <105 mmHg and with >15 mmHg increase from baseline: Week 4: number analyzed (Participants) | 44 | 50
  DBP (mmHg): <105 mmHg and with >15 mmHg increase from baseline: Week 4 | 0 | 0
  Temperature (degree C): <35.5 degree C: Week 4: number analyzed (Participants) | 44 | 50
  Temperature (degree C): <35.5 degree C: Week 4 | 0 | 0
  Temperature (degree C): >37.5 degree C: Week 4: number analyzed (Participants) | 44 | 50
  Temperature (degree C): >37.5 degree C: Week 4 | 0 | 0
  Respiratory Rate: >20 breaths per minute: Week 4: number analyzed (Participants) | 44 | 50
  Respiratory Rate: >20 breaths per minute: Week 4 | 0 | 0
  Pulse: <50 bpm and with >15 bpm decrease from baseline: Week 6: number analyzed (Participants) | 42 | 50
  Pulse: <50 bpm and with >15 bpm decrease from baseline: Week 6 | 0 | 0
  Pulse: <100 bpm and with >15 bpm increase from baseline: Week 6: number analyzed (Participants) | 42 | 50
  Pulse: <100 bpm and with >15 bpm increase from baseline: Week 6 | 0 | 0
  SBP (mmHg): <90 mmHg and with >20 mmHg decrease from baseline: Week 6: number analyzed (Participants) | 42 | 50
  SBP (mmHg): <90 mmHg and with >20 mmHg decrease from baseline: Week 6 | 0 | 0
  SBP (mmHg): >180 mmHg and with >20 mmHg increase from baseline: Week 6: number analyzed (Participants) | 42 | 50
  SBP (mmHg): >180 mmHg and with >20 mmHg increase from baseline: Week 6 | 0 | 0
  DBP (mmHg): <50 mmHg and with >15 mmHg decrease from baseline: Week 6: number analyzed (Participants) | 42 | 50
  DBP (mmHg): <50 mmHg and with >15 mmHg decrease from baseline: Week 6 | 0 | 0
  DBP (mmHg): >105 mmHg and with >15 mmHg increase from baseline: Week 6: number analyzed (Participants) | 42 | 50
  DBP (mmHg): >105 mmHg and with >15 mmHg increase from baseline: Week 6 | 0 | 0
  Temperature (C): <35.5 degree C: Week 6: number analyzed (Participants) | 42 | 50
  Temperature (C): <35.5 degree C: Week 6 | 0 | 0
  Temperature (degree C): <37.5 degree C: Week 6: number analyzed (Participants) | 42 | 50
  Temperature (degree C): <37.5 degree C: Week 6 | 0 | 0
  Respiratory Rate (breaths/min): >20 breaths per minute: Week 6: number analyzed (Participants) | 42 | 50
  Respiratory Rate (breaths/min): >20 breaths per minute: Week 6 | 0 | 0
  Weight (kg): Decrease from baseline >7%: Week 6: number analyzed (Participants) | 42 | 50
  Weight (kg): Decrease from baseline >7%: Week 6 | 0 | 0
  Weight (kg): Increase from baseline >7%: Week 6: number analyzed (Participants) | 42 | 50
  Weight (kg): Increase from baseline >7%: Week 6 | 0 | 1
  Pulse: <50 bpm and with >15 bpm decrease from baseline: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  Pulse: <50 bpm and with >15 bpm decrease from baseline: Follow-up (Week 8) | 0 | 0
  Pulse: >100 bpm and with >15 bpm increase from baseline: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  Pulse: >100 bpm and with >15 bpm increase from baseline: Follow-up (Week 8) | 1 | 0
  SBP (mmHg): <90mmHg and with >20 mmHg decrease from baseline: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  SBP (mmHg): <90mmHg and with >20 mmHg decrease from baseline: Follow-up (Week 8) | 0 | 0
  SBP (mmHg):>180mmHg and with >20 mmHg increase from baseline: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  SBP (mmHg):>180mmHg and with >20 mmHg increase from baseline: Follow-up (Week 8) | 0 | 1
  DBP (mmHg): <50mmHg and with >15mmHg decrease from baseline: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  DBP (mmHg): <50mmHg and with >15mmHg decrease from baseline: Follow-up (Week 8) | 0 | 0
  DBP (mmHg):>105mmHg and with >15mmHg increase from baseline: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  DBP (mmHg):>105mmHg and with >15mmHg increase from baseline: Follow-up (Week 8) | 0 | 1
  Temperature (C): <35.5 degree C: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  Temperature (C): <35.5 degree C: Follow-up (Week 8) | 0 | 0
  Temperature (C): >37.5 degree C: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  Temperature (C): >37.5 degree C: Follow-up (Week 8) | 0 | 0
  Respiratory Rate (breaths/min): >20 breaths per minute: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  Respiratory Rate (breaths/min): >20 breaths per minute: Follow-up (Week 8) | 0 | 0
  Weight (kg): Decrease from baseline >7%: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  Weight (kg): Decrease from baseline >7%: Follow-up (Week 8) | 1 | 0
  Weight (kg): Increase from baseline >7%: Follow-up (Week 8): number analyzed (Participants) | 42 | 48
  Weight (kg): Increase from baseline >7%: Follow-up (Week 8) | 0 | 2

7. Secondary Outcome: Change From Baseline in Clinical Laboratory Values in Male Hormone: Inhibin B
Description: Change from baseline in clinical laboratory values in male hormone (Inhibin B) were reported.
Time Frame: Baseline (Day 1), Week 4, 6, and 8 (Follow-up/Early Withdrawal)
Population: Safety analysis set included all randomized participants who took at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed at specified timepoints.
Measure: Mean (Standard Deviation); unit: nanograms per liter (ng/L)
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 16 | 25
nanograms per liter (ng/L)
  Week 4: number analyzed (Participants) | 15 | 22
  Week 4 | -5.9 (30.45) | 3.1 (22.15)
  Week 6: number analyzed (Participants) | 14 | 21
  Week 6 | -2.1 (30.02) | -1.8 (31.09)
  Week 8: number analyzed (Participants) | 14 | 21
  Week 8 | -1.2 (28.25) | 7.3 (19.60)

8. Secondary Outcome: Change From Baseline in Clinical Laboratory Values in Male Hormone: Luteinizing Hormone
Description: Change from baseline in clinical laboratory values in male hormone (luteinizing hormone) were reported.
Time Frame: Baseline (Day 1), Week 4, 6, and 8 (Follow-up/Early Withdrawal)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: International units per liter (IU/L)
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 16 | 27
International units per liter (IU/L)
  Week 4: number analyzed (Participants) | 15 | 24
  Week 4 | 0.15 (1.814) | 0.29 (1.513)
  Week 6: number analyzed (Participants) | 16 | 24
  Week 6 | -0.11 (1.677) | 0.63 (2.719)
  Week 8 | -0.35 (1.638) | 0.84 (2.103)

9. Secondary Outcome: Change From Baseline in Clinical Laboratory Values in Male Hormone: Prolactin
Description: Change from baseline in clinical laboratory values in male hormone (prolactin) were reported.
Time Frame: Baseline (Day 1), Week 4, 6, and 8 (Follow-up/Early Withdrawal)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: micrograms per liter (mcg/L)
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 16 | 27
micrograms per liter (mcg/L)
  Week 4: number analyzed (Participants) | 15 | 24
  Week 4 | 0.347 (2.4360) | 1.803 (3.6211)
  Week 6: number analyzed (Participants) | 16 | 24
  Week 6 | 0.551 (3.1575) | 1.465 (5.3742)
  Week 8 | -0.160 (3.8622) | 1.748 (3.9231)

10. Secondary Outcome: Change From Baseline in Clinical Laboratory Values in Male Hormones: Sex Hormone Binding Globulin, Testosterone (Free), Testosterone (High Sensitivity), and Testosterone (Low Sensitivity)
Description: Change from baseline in clinical laboratory values in male hormones (sex hormone binding globulin, testosterone [free], testosterone [high sensitivity], and testosterone [low sensitivity]) were reported.
Time Frame: Baseline (Day 1), Week 4, 6, and 8 (Follow-up/Early Withdrawal)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanomoles per liter (nmol/L)
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 16 | 27
nanomoles per liter (nmol/L)
  Sex Hormone Binding Globulin: Week 4: number analyzed (Participants) | 15 | 23
  Sex Hormone Binding Globulin: Week 4 | -1.976 (7.1297) | -0.574 (8.5796)
  Sex Hormone Binding Globulin: Week 6: number analyzed (Participants) | 16 | 23
  Sex Hormone Binding Globulin: Week 6 | -4.020 (7.4992) | -0.274 (9.2454)
  Sex Hormone Binding Globulin: Week 8 | -2.520 (7.8489) | 1.058 (6.6109)
  Testosterone, Free: Week 4: number analyzed (Participants) | 12 | 15
  Testosterone, Free: Week 4 | 0.005 (0.0677) | 0.030 (0.0995)
  Testosterone, Free: Week 6: number analyzed (Participants) | 13 | 18
  Testosterone, Free: Week 6 | -0.010 (0.0731) | 0.037 (0.1084)
  Testosterone, Free: Week 8: number analyzed (Participants) | 13 | 16
  Testosterone, Free: Week 8 | 0.031 (0.0763) | 0.046 (0.0877)
  Testosterone, High Sensitivity: Week 4 | -0.797 (3.3271) | 0.357 (5.5917)
  Testosterone, High Sensitivity: Week 6 | -1.262 (3.6807) | 0.842 (5.6815)
  Testosterone, High Sensitivity: Week 8 | 0.604 (3.7718) | 1.416 (4.3083)
  Testosterone, Low Sensitivity: Week 4 | -0.791 (3.8886) | 0.854 (5.9616)
  Testosterone, Low Sensitivity: Week 6 | -1.532 (4.5203) | 1.380 (5.9515)
  Testosterone, Low Sensitivity: Week 8 | 1.116 (4.8452) | 1.728 (4.6578)

11. Secondary Outcome: Number of Participants With Abnormal Laboratory Values: Serum Chemistry
Description: Number of participants with abnormal laboratory values: serum chemistry were reported. It included: aspartate aminotransferase (high), alanine aminotransferase (high), bilirubin (high/low), and alkaline phosphatase (high/low). Only categories with data were reported.
Time Frame: Weeks 2, 4, 6, and 8 (Follow-up/Early Withdrawal)
Population: Safety analysis set included all randomized participants who took at least 1 dose of study intervention. Here, 'n' (number analyzed) is defined as participants analyzed at specified categories.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 54 | 60
Participants
  Aspartate Aminotransferase (High): Week 2: number analyzed (Participants) | 44 | 55
  Aspartate Aminotransferase (High): Week 2 | 2 | 2
  Aspartate Aminotransferase (High): Week 4: number analyzed (Participants) | 43 | 50
  Aspartate Aminotransferase (High): Week 4 | 0 | 2
  Aspartate Aminotransferase (High): Week 6: number analyzed (Participants) | 42 | 49
  Aspartate Aminotransferase (High): Week 6 | 1 | 0
  Aspartate Aminotransferase (High): Week 8: number analyzed (Participants) | 54 | 50
  Aspartate Aminotransferase (High): Week 8 | 0 | 2
  Alanine Aminotransferase (High): Week 2: number analyzed (Participants) | 45 | 60
  Alanine Aminotransferase (High): Week 2 | 1 | 3
  Alanine Aminotransferase (High): Week 4: number analyzed (Participants) | 42 | 50
  Alanine Aminotransferase (High): Week 4 | 2 | 3
  Alanine Aminotransferase (High): Week 6: number analyzed (Participants) | 41 | 49
  Alanine Aminotransferase (High): Week 6 | 2 | 1
  Alanine Aminotransferase (High): Week 8: number analyzed (Participants) | 54 | 49
  Alanine Aminotransferase (High): Week 8 | 1 | 2
  Bilirubin (Low): Week 2: number analyzed (Participants) | 45 | 60
  Bilirubin (Low): Week 2 | 4 | 9
  Bilirubin (High): Week 2: number analyzed (Participants) | 45 | 60
  Bilirubin (High): Week 2 | 1 | 0
  Bilirubin (Low): Week 4: number analyzed (Participants) | 43 | 50
  Bilirubin (Low): Week 4 | 8 | 7
  Bilirubin (Low): Week 6: number analyzed (Participants) | 42 | 50
  Bilirubin (Low): Week 6 | 5 | 4
  Bilirubin (High): Week 6: number analyzed (Participants) | 42 | 50
  Bilirubin (High): Week 6 | 2 | 0
  Bilirubin (Low): Week 8: number analyzed (Participants) | 54 | 50
  Bilirubin (Low): Week 8 | 3 | 5
  Bilirubin (High): Week 8: number analyzed (Participants) | 54 | 50
  Bilirubin (High): Week 8 | 1 | 0
  Alkaline Phosphatase (Low): Week 2: number analyzed (Participants) | 45 | 60
  Alkaline Phosphatase (Low): Week 2 | 1 | 0
  Alkaline Phosphatase (High): Week 2: number analyzed (Participants) | 45 | 60
  Alkaline Phosphatase (High): Week 2 | 3 | 5
  Alkaline Phosphatase (Low): Week 4: number analyzed (Participants) | 42 | 50
  Alkaline Phosphatase (Low): Week 4 | 1 | 0
  Alkaline Phosphatase (High): Week 4: number analyzed (Participants) | 42 | 50
  Alkaline Phosphatase (High): Week 4 | 0 | 3
  Alkaline Phosphatase (Low): Week 6: number analyzed (Participants) | 42 | 49
  Alkaline Phosphatase (Low): Week 6 | 1 | 0
  Alkaline Phosphatase (High): Week 6: number analyzed (Participants) | 42 | 49
  Alkaline Phosphatase (High): Week 6 | 1 | 6
  Alkaline Phosphatase (Low): Week 8: number analyzed (Participants) | 54 | 50
  Alkaline Phosphatase (Low): Week 8 | 1 | 0
  Alkaline Phosphatase (High): Week 8: number analyzed (Participants) | 54 | 50
  Alkaline Phosphatase (High): Week 8 | 4 | 5

12. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values: Hematology
Description: Number of participants with clinically significant abnormal laboratory values: hematology were reported.
Time Frame: Weeks 2, 4, 6, and 8 (Follow-up/Early Withdrawal)
Population: Safety analysis set included all randomized participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 54 | 60
Participants
  Week 2 | 0 | 0
  Week 4 | 0 | 0
  Week 6 | 0 | 0
  Week 8 | 0 | 0

13. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Laboratory Values: Urinalysis
Description: Number of participants with clinically significant abnormal laboratory values: urinalysis were reported.
Time Frame: Weeks 2, 4, 6, and 8 (Follow-up/Early Withdrawal)
Population: Safety analysis set included all randomized participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 54 | 60
Participants
  Week 2 | 0 | 0
  Week 4 | 0 | 0
  Week 6 | 0 | 0
  Week 8 | 0 | 0

14. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs were reported. An adverse event (AE) is any untoward medical occurrence in a clinical study participants who administered a medicinal (investigational or non-investigational) product and does not necessarily have a causal relationship with the treatment. A TEAE defined as an AE that occurred at or after the first dose administration up to day of the last dose plus 30 days.
Time Frame: Day 1 (Week 0) up to 30 days after the last dose (up to 11 weeks)
Population: Safety analysis set included all randomized participants who took at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 54 | 60
Participants | 22 | 28

15. Secondary Outcome: Number of Participants With Treatment-emergent Abnormalities in Electrocardiograms (ECGs)
Description: Number of participants with treatment-emergent abnormalities in ECGs were reported. It included ECG mean heart rate (abnormally low [AL]: <50 and abnormally high [AH]: >100 beats per minute [bpm]), PR Interval (AL: <120 and AH: >200 milliseconds [msec]), QRS Duration (AL: <60 and AH: >120 msec), and QT Interval (AL: <200 and AH: >500 msec). A treatment-emergent abnormalities in ECGs are defined as those abnormalities that occurred at or after the first dose administration.
Time Frame: Weeks 1, 2, 4, 6, and 8 (Follow-up/Early Withdrawal)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 54 | 60
Participants
  ECG Mean Heart Rate: <50 bpm: Week 1: number analyzed (Participants) | 48 | 60
  ECG Mean Heart Rate: <50 bpm: Week 1 | 1 | 0
  ECG Mean Heart Rate: >100 bpm: Week 1: number analyzed (Participants) | 48 | 60
  ECG Mean Heart Rate: >100 bpm: Week 1 | 0 | 0
  PR Interval: <120 msec: Week 1: number analyzed (Participants) | 48 | 60
  PR Interval: <120 msec: Week 1 | 0 | 1
  PR Interval: >200 msec: Week 1: number analyzed (Participants) | 48 | 60
  PR Interval: >200 msec: Week 1 | 1 | 0
  QRS Duration: <60 msec: Week 1: number analyzed (Participants) | 48 | 60
  QRS Duration: <60 msec: Week 1 | 0 | 1
  QRS Duration: >120 msec: Week 1: number analyzed (Participants) | 48 | 60
  QRS Duration: >120 msec: Week 1 | 1 | 0
  QT Interval: <200 msec: Week 1: number analyzed (Participants) | 48 | 60
  QT Interval: <200 msec: Week 1 | 0 | 0
  QT Interval: >500 msec: Week 1: number analyzed (Participants) | 48 | 60
  QT Interval: >500 msec: Week 1 | 0 | 0
  ECG Mean Heart Rate: <50 bpm: Week 2: number analyzed (Participants) | 44 | 60
  ECG Mean Heart Rate: <50 bpm: Week 2 | 0 | 0
  ECG Mean Heart Rate: >100 bpm: Week 2: number analyzed (Participants) | 44 | 60
  ECG Mean Heart Rate: >100 bpm: Week 2 | 1 | 1
  PR Interval: <120 msec: Week 2: number analyzed (Participants) | 44 | 60
  PR Interval: <120 msec: Week 2 | 0 | 0
  PR Interval: >200 msec: Week 2: number analyzed (Participants) | 44 | 60
  PR Interval: >200 msec: Week 2 | 1 | 2
  QRS Duration: <60 msec: Week 2: number analyzed (Participants) | 44 | 60
  QRS Duration: <60 msec: Week 2 | 0 | 1
  QRS Duration: >120 msec: Week 2: number analyzed (Participants) | 44 | 60
  QRS Duration: >120 msec: Week 2 | 0 | 1
  QT Interval: <200 msec: Week 2: number analyzed (Participants) | 44 | 60
  QT Interval: <200 msec: Week 2 | 0 | 0
  QT Interval: >500 msec: Week 2: number analyzed (Participants) | 44 | 60
  QT Interval: >500 msec: Week 2 | 0 | 0
  ECG Mean Heart Rate: <50 bpm: Week 4: number analyzed (Participants) | 44 | 50
  ECG Mean Heart Rate: <50 bpm: Week 4 | 0 | 0
  ECG Mean Heart Rate: >100 bpm: Week 4: number analyzed (Participants) | 44 | 50
  ECG Mean Heart Rate: >100 bpm: Week 4 | 1 | 0
  PR Interval: <120 msec: Week 4: number analyzed (Participants) | 44 | 50
  PR Interval: <120 msec: Week 4 | 0 | 1
  PR Interval: >200 msec: Week 4: number analyzed (Participants) | 44 | 50
  PR Interval: >200 msec: Week 4 | 0 | 0
  QRS Duration: <60 msec: Week 4: number analyzed (Participants) | 44 | 50
  QRS Duration: <60 msec: Week 4 | 0 | 1
  QRS Duration: >120 msec: Week 4: number analyzed (Participants) | 44 | 50
  QRS Duration: >120 msec: Week 4 | 1 | 0
  QT Interval: <200 msec: Week 4: number analyzed (Participants) | 44 | 50
  QT Interval: <200 msec: Week 4 | 0 | 0
  QT Interval: >500 msec: Week 4: number analyzed (Participants) | 44 | 50
  QT Interval: >500 msec: Week 4 | 0 | 0
  ECG Mean Heart Rate: <50 bpm: Week 6: number analyzed (Participants) | 41 | 50
  ECG Mean Heart Rate: <50 bpm: Week 6 | 0 | 0
  ECG Mean Heart Rate: >100 bpm: Week 6: number analyzed (Participants) | 41 | 50
  ECG Mean Heart Rate: >100 bpm: Week 6 | 0 | 0
  PR Interval: <120 msec: Week 6: number analyzed (Participants) | 41 | 50
  PR Interval: <120 msec: Week 6 | 0 | 0
  PR Interval: >200 msec: Week 6: number analyzed (Participants) | 41 | 50
  PR Interval: >200 msec: Week 6 | 0 | 0
  QRS Duration: <60 msec: Week 6: number analyzed (Participants) | 41 | 50
  QRS Duration: <60 msec: Week 6 | 0 | 4
  QRS Duration: >120 msec: Week 6: number analyzed (Participants) | 41 | 50
  QRS Duration: >120 msec: Week 6 | 0 | 0
  QT Interval: <200 msec: Week 6: number analyzed (Participants) | 41 | 50
  QT Interval: <200 msec: Week 6 | 0 | 0
  QT Interval: >500 msec: Week 6: number analyzed (Participants) | 41 | 50
  QT Interval: >500 msec: Week 6 | 0 | 0
  ECG Mean Heart Rate: <50 bpm: Week 8: number analyzed (Participants) | 54 | 52
  ECG Mean Heart Rate: <50 bpm: Week 8 | 0 | 0
  ECG Mean Heart Rate: >100 bpm: Week 8: number analyzed (Participants) | 54 | 52
  ECG Mean Heart Rate: >100 bpm: Week 8 | 0 | 0
  PR Interval: <120 msec: Week 8: number analyzed (Participants) | 54 | 52
  PR Interval: <120 msec: Week 8 | 1 | 0
  PR Interval: >200 msec: Week 8: number analyzed (Participants) | 54 | 52
  PR Interval: >200 msec: Week 8 | 0 | 0
  QRS Duration: <60 msec: Week 8: number analyzed (Participants) | 54 | 52
  QRS Duration: <60 msec: Week 8 | 1 | 2
  QRS Duration: >120 msec: Week 8: number analyzed (Participants) | 54 | 52
  QRS Duration: >120 msec: Week 8 | 0 | 1
  QT Interval: <200 msec: Week 8: number analyzed (Participants) | 54 | 52
  QT Interval: <200 msec: Week 8 | 0 | 0
  QT Interval: >500 msec: Week 8: number analyzed (Participants) | 54 | 52
  QT Interval: >500 msec: Week 8 | 0 | 0

16. Secondary Outcome: Change From Baseline in Young Mania Rating Scale (YMRS) Total Score
Description: Change from baseline in YMRS total score were reported. The YMRS was designed to measure the severity of manic symptoms, to gauge the effect of treatment on mania severity, and to detect a return of manic symptoms (for example relapse or recurrence). YMRS had 11 items : 4 items (irritability, speech, thought content, and disruptive/aggressive behavior) were graded on a scale of 0 to 8 and the remaining 7 items (elevated mood, increased motor activity, sexual interest, sleep, language-thought disorder, appearance, and insight) were graded on a scale of 0 to 4. Higher scores indicated greater symptom severity. Responses were summed to yield YMRS total score ranged from 0 to 60 , with higher scores reflecting greater severity of mania.
Time Frame: From Baseline (Day 1) up to Week 6
Population: Safety analysis set included all randomized participants who took at least 1 dose of study intervention. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 42 | 50
Units on a scale | -1.2 (2.23) | -1.1 (1.81)

17. Secondary Outcome: Number of Participants Who Reported Suicidal Ideation (SI) or Suicidal Behavior (SB) Using With Columbia Suicide Severity Rating Scale (C-SSRS) Score
Description: C-SSRS is a clinician-rated instrument that reports severity of both suicidal ideation (SI) and suicidal behavior (SB). SI categories: 1 (wish to be dead), 2 (nonspecific active suicidal thoughts), 3 (active suicidal ideation with any methods [not plan] without intent to act), 4 (active SI with some intent to act, without specific plan), and 5 (active SI with specific plan and intent). SB categories: 6 (preparatory acts or behavior), 7 (aborted attempt), 8 (interrupted attempt), 9 (actual attempt), and 10 (suicide). An additional category for non-suicide: non-suicidal self-injurious behavior. SI/SB was indicated by a "yes" answer to any of the listed categories. Score of 0 (no SI or SB) was assigned. Maximum score of 1 to 10 was assigned if suicidal ideation or behavior was present. Scoring was grouped into 3 categories: No SI/SB (0), SI (score 1 to 5), and SB (score 6 to 10), with higher scores indicating more severe ideation/behavior.
Time Frame: From Baseline (Day 1) up to Week 8
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 53 | 59
Participants
  Suicidal ideation | 3 | 6
  Suicidal behavior | 1 | 0
  No SI/SB | 49 [lower limit 2.23] | 53 [lower limit 1.81]

18. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity Scale (CGI-S) Score
Description: Change from baseline in CGI-S score were reported. The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness that takes into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S is a 7-point global assessment scale that measures the clinician's impression of the severity of mental illness exhibited by a participant, and rated on a scale of 1 to 7: 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; and 7=among the most extremely ill participants. Higher scores indicate worsening. Negative change in CGI-S score indicate improvement.
Time Frame: From Baseline (Day 1) up to Week 6
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 42 | 50
Units on a scale | -1.9 (1.49) | -1.7 (1.32)

19. Secondary Outcome: Plasma Concentrations of JNJ-55308942
Description: Plasma concentrations of JNJ-55308942 were reported.
Time Frame: Predose, 1.5 hours and 4 hours post-dose on Week 0 (Day 1), Weeks 1 (Day 8), 2 (Day 15), 4 (Day 29), and 6 (Day 43)
Population: Pharmacokinetics (PK) analysis set included all participants who received at least 1 dose of JNJ-55308942 and had at least 1 valid blood sample drawn for PK analysis. Here, 'n' (number analyzed) is defined as participants analyzed at specified categories. Data for this outcome measure was not planned to be collected and analyzed for placebo arm.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | JNJ-55308942
Number analyzed (Participants) | 53
Nanograms per milliliter (ng/mL)
  Week 0 (Day 1): Predose: number analyzed (Participants) | 51
  Week 0 (Day 1): Predose | 0.00 (0.000)
  Week 0 (Day 1): 1.5 hours postdose | 406.13 (162.407)
  Week 0 (Day 1): 4 hours postdose: number analyzed (Participants) | 49
  Week 0 (Day 1): 4 hours postdose | 407.72 (133.461)
  Week 1 (Day 8): Predose: number analyzed (Participants) | 46
  Week 1 (Day 8): Predose | 531.20 (200.351)
  Week 1 (Day 8): 1.5 hours postdose: number analyzed (Participants) | 46
  Week 1 (Day 8): 1.5 hours postdose | 868.01 (296.255)
  Week 1 (Day 8): 4 hours postdose: number analyzed (Participants) | 46
  Week 1 (Day 8): 4 hours postdose | 892.54 (219.210)
  Week 2 (Day 15): Predose: number analyzed (Participants) | 44
  Week 2 (Day 15): Predose | 561.32 (194.184)
  Week 2 (Day 15): 1.5 hours postdose: number analyzed (Participants) | 44
  Week 2 (Day 15): 1.5 hours postdose | 930.59 (265.581)
  Week 2 (Day 15): 4 hours postdose: number analyzed (Participants) | 44
  Week 2 (Day 15): 4 hours postdose | 919.86 (213.028)
  Week 4 (Day 29): Predose: number analyzed (Participants) | 42
  Week 4 (Day 29): Predose | 528.90 (144.580)
  Week 4 (Day 29): 1.5 hours postdose: number analyzed (Participants) | 44
  Week 4 (Day 29): 1.5 hours postdose | 885.50 (249.562)
  Week 4 (Day 29): 4 hours postdose: number analyzed (Participants) | 44
  Week 4 (Day 29): 4 hours postdose | 872.80 (208.734)
  Week 6 (Day 43): Predose: number analyzed (Participants) | 41
  Week 6 (Day 43): Predose | 535.80 (160.568)
  Week 6 (Day 43): 1.5 hours postdose: number analyzed (Participants) | 39
  Week 6 (Day 43): 1.5 hours postdose | 862.31 (240.540)
  Week 6 (Day 43): 4 hours postdose: number analyzed (Participants) | 41
  Week 6 (Day 43): 4 hours postdose | 883.51 (209.413)

20. Secondary Outcome: Change From Baseline in Patient Reported Outcomes Measurement Information System (PROMIS) Score - Ability to Participate in Social Roles and Activities (APS) T-Scores
Description: Change from baseline in PROMIS score - ability to participate in social roles and activities T-Scores were reported. The PROMIS - APS item bank assessed the perceived ability to perform one's usual social roles and activities. The item bank did not use a time frame (for example, over the past seven days) when assessing the APS. The Short Form 4a included 4 items that represent this concept. Each question had 5 response options ranging in value from 1 to 5 with higher scores indicating better social function. The total raw score for the short form was calculated by summing the values of the response to each question, so for the 4-item form, the lowest possible raw score was 4; the highest possible raw score was 20. The total raw score was converted to a T score with a mean of 50 and a standard deviation of 10. Higher T-scores indicate better social function.
Time Frame: Baseline (Day 1), Weeks 1, 2, 3, 4, 5, and 6
Population: FAS included all randomized participants who received at least 1 dose of study intervention and had both the baseline and at least 1 postbaseline MADRS measurement. Here, 'n' (number analyzed) is defined as participants analyzed at specified categories.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 48 | 59
T-score
  PROMIS-APS T-score: Week 1: number analyzed (Participants) | 48 | 57
  PROMIS-APS T-score: Week 1 | 2.51 (5.682) | 1.69 (6.859)
  PROMIS-APS T-score: Week 2: number analyzed (Participants) | 45 | 56
  PROMIS-APS T-score: Week 2 | 5.33 (6.901) | 4.49 (9.174)
  PROMIS-APS T-score: Week 3: number analyzed (Participants) | 42 | 52
  PROMIS-APS T-score: Week 3 | 6.52 (8.226) | 5.00 (8.884)
  PROMIS-APS T-score: Week 4: number analyzed (Participants) | 43 | 49
  PROMIS-APS T-score: Week 4 | 9.12 (9.018) | 6.07 (8.369)
  PROMIS-APS T-score: Week 5: number analyzed (Participants) | 41 | 47
  PROMIS-APS T-score: Week 5 | 9.47 (8.248) | 4.90 (9.296)
  PROMIS-APS T-score: Week 6: number analyzed (Participants) | 42 | 50
  PROMIS-APS T-score: Week 6 | 10.50 (8.211) | 6.12 (8.412)

21. Secondary Outcome: Change From Baseline in Patient Health Questionnaire-9 (PHQ-9) Total Score
Description: Change from baseline in PHQ-9 total score were reported. PHQ-9 is 9-item, self-report scale assessed depressive symptoms. Each item was rated on 4-point scale (0=Not at all, 1=several days, 2=more than half days, 3=nearly every day. The participant's item responses were summed to provide PHQ-9 total score (range of 0 to 27) with higher scores indicating greater severity of depressive symptoms.
Time Frame: Baseline (Day 1), Weeks 1, 2, 3, 4, 5, and 6
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 48 | 59
Units on a scale
  Week 1: number analyzed (Participants) | 48 | 57
  Week 1 | -2.8 (4.24) | -3.1 (5.45)
  Week 2: number analyzed (Participants) | 45 | 56
  Week 2 | -5.2 (5.64) | -4.7 (6.63)
  Week 3: number analyzed (Participants) | 41 | 52
  Week 3 | -6.4 (6.25) | -5.1 (6.90)
  Week 4: number analyzed (Participants) | 43 | 49
  Week 4 | -7.0 (6.38) | -6.1 (6.81)
  Week 5: number analyzed (Participants) | 41 | 47
  Week 5 | -8.2 (6.59) | -5.2 (7.21)
  Week 6: number analyzed (Participants) | 42 | 50
  Week 6 | -9.0 (6.79) | -7.0 (7.41)

22. Secondary Outcome: Change From Baseline in Generalized Anxiety Disorder 7 (GAD-7) Total Score
Description: Change from baseline in GAD-7 total score were reported. GAD-7 is a brief and validated 7-item self-reported questionnaire for assessment of overall GAD. Participants responded to each item using a 4-point scale with response categories of 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day, with a higher score representing a more severe condition. Item responses were summed to yield GAD-7 total score which ranged of 0 to 21, where higher scores indicated more anxiety.
Time Frame: Baseline (Day 1), Weeks 2, 4, and 6
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 48 | 59
Units on a scale
  Week 2: number analyzed (Participants) | 45 | 56
  Week 2 | -3.8 (5.08) | -4.2 (5.76)
  Week 4: number analyzed (Participants) | 44 | 50
  Week 4 | -5.0 (6.59) | -4.5 (5.14)
  Week 6: number analyzed (Participants) | 42 | 50
  Week 6 | -5.7 (6.21) | -5.7 (5.77)

23. Secondary Outcome: Number of Participants Who Achieved Response at Week 6
Description: Number of participants who achieved response at Week 6 were reported. Response was defined as greater than or equal to (>=)50% improvement in MADRS total score from baseline. MADRS was a clinician-rated scale designed to measure depression severity and detect changes due to AD treatment. The MADRS evaluated reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The scale consisted of 10 items, each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms),with higher score indicating a more severe condition. The MADRS total score was the sum of scores from individual question items and it ranged from 0 to 60, with higher scores indicated more severe conditions. Negative change in MADRS total score indicated improvement.
Time Frame: Week 6
Population: FAS included all randomized participants who received at least 1 dose of study intervention and have both the baseline and at least 1 postbaseline MADRS measurement.
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 48 | 59
Participants | 27 [lower limit 6.21] | 31 [lower limit 5.77]

24. Secondary Outcome: Number of Participants Who Achieved Remission at Week 6
Description: Number of participants who achieved remission at Week 6 were reported. Remission was defined as MADRS total score <=12. MADRS was a clinician-rated scale designed to measure depression severity and detect changes due to AD treatment. The MADRS evaluated reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The scale consisted of 10 items, each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms),with higher score indicating a more severe condition. The MADRS total score was the sum of scores from individual question items and it ranged from 0 to 60, with higher scores indicated more severe conditions. Negative change in MADRS total score indicated improvement.
Time Frame: Week 6
Population: as for outcome 23
Measure: Count of Participants; unit: Participants
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 48 | 59
Participants | 25 [lower limit 6.21] | 30 [lower limit 5.77]

25. Secondary Outcome: Change From Baseline in MADRS Total Score up to Week 6 (Subgroup of Participants With Messenger Ribonucleic Acid [mRNA] Transcript Levels)
Description: Change from baseline in MADRS total score up to Week 6 (subgroup of participants with mRNA transcript levels) was planned to be reported. Subgroup included participants with mRNA transcript levels at baseline that exceeded the medium level for both P2RX7 and IL-1-beta. MADRS was a clinician-rated scale designed to measure depression severity and detect changes due to AD treatment. MADRS evaluated reported sadness, apparent sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, and suicidal thoughts. The scale consisted of 10 items, each of which was scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms),with higher score indicating a more severe condition. MADRS total score was the sum of scores from individual question items and it ranged from 0 to 60, with higher scores indicated more severe conditions. Negative change in MADRS total score indicated improvement.
Time Frame: From Baseline (Day 1) up to Week 6
Population: FAS included all randomized participants who had received at least 1 dose of study intervention and have both the baseline and at least 1 postbaseline MADRS measurement.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 48 | 59
Units on a scale | NA (NA) — NA refers that mean and standard deviation were not calculable under acceptable margins for categorization of participants because of poor reproducibility of the PCR method using small RNA volumes, participants could not be categorized by mRNA transcript levels. | NA (NA) — NA refers that mean and standard deviation were not calculable under acceptable margins for categorization of participants because of poor reproducibility of the PCR method using small RNA volumes, participants could not be categorized by mRNA transcript levels.

26. Secondary Outcome: Change From Baseline in MADRS Total Score up to Week 6 (Concomitant Medication Subgroup Analysis)
Description: Change from baseline in MADRS total score up to Week 6 (concomitant medication subgroup analysis) was reported. Concomitant medication subgroup analysis included subjects with BD not taking any mood stabilizer or antipsychotic, taking a mood stabilizer alone, taking antipsychotic alone, and taking a combination of mood stabilizer and an antipsychotic. MADRS measures depression severity, detects changes due to AD treatment. It consists of 10 items (evaluate apparent sadness, reported sadness, inner tension, reduced sleep, reduced appetite, concentration difficulties, lassitude, inability to feel, pessimistic thoughts, suicidal thoughts), scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed to total possible score of 0 to 60. Higher scores indicate more severe conditions. Negative change in score indicates improvement.
Time Frame: From Baseline (Day 1) up to Week 6
Population: FAS included all randomized participants who had received at least 1 dose of study intervention and have both the baseline and at least 1 postbaseline MADRS measurement. Here, 'N' (overall number of participants analyzed) signifies number of participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed at specified categories. n=0 signifies no participant was available for the analysis.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | JNJ-55308942 | Placebo
Number analyzed (Participants) | 42 | 50
Units on a scale
  Concomitant medication status: Not taking any mood stabilizer or antipsychotic: number analyzed (Participants) | 11 | 19
  Concomitant medication status: Not taking any mood stabilizer or antipsychotic | -15.5 (13.18) | -16.2 (9.69)
  Concomitant medication status: Taking a mood stabilizer alone: number analyzed (Participants) | 29 | 30
  Concomitant medication status: Taking a mood stabilizer alone | -16.3 (9.82) | -15.6 (9.47)
  Concomitant medication status: Taking an antipsychotic alone: number analyzed (Participants) | 1 | 1
  Concomitant medication status: Taking an antipsychotic alone | -13.0 (NA) — NA refers to standard deviation was not estimable as only 1 participant was analyzed. | 5.0 (NA) — NA refers to standard deviation was not estimable as only 1 participant was analyzed.
  Concomitant medication status: Taking a combination of a mood stabilizer and an antipsychotic: number analyzed (Participants) | 1 | 0
  Concomitant medication status: Taking a combination of a mood stabilizer and an antipsychotic | -13.0 (NA) — NA refers to standard deviation was not estimable as only 1 participant was analyzed. |

ADVERSE EVENTS:
Time Frame: All-cause mortality: From screening (-28 days) up to end of study (up to 12 weeks); SAEs and Other AEs: From Day 1 (Week 0) up to 30 days after the last dose (up to 11 weeks)
Description: All-cause mortality was analyzed on all randomized participants in the study. SAEs and Other AEs were analyzed on safety analysis set that included all randomized participants who took at least 1 dose of study intervention.
Arm/Group | JNJ-55308942 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/61
Serious Adverse Events (participants affected / at risk) | 2/54 | 3/60
Other Adverse Events (participants affected / at risk) | 6/54 | 10/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-55308942 (N=54) | Placebo (N=60)
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 0 | 1
Behaviour Disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JNJ-55308942 (N=54) | Placebo (N=60)
Diarrhoea (Gastrointestinal disorders) | 2 | 3
Nausea (Gastrointestinal disorders) | 4 | 5
Vomiting (Gastrointestinal disorders) | 1 | 3
Headache (Nervous system disorders) | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT05328297/Prot_000.pdf
  • Statistical Analysis Plan (2024-06-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05328297/SAP_001.pdf